CLINICAL TRIAL: NCT07090876
Title: Hemodynamic Effects of a Standardized Grape Seed Extract Supplementation: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Clinical Trial
Brief Title: Hemodynamic Effects of a Standardized Grape Seed Extract Supplementation
Acronym: ZENITH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indena S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZENITH_RCT2025
Record Dates: First submitted 2025-07-17; First posted 2025-07-29 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-07

CONDITIONS: High-normal Blood Pressure
Keywords: High-normal blood pressure; Grape seed extract; Dietary supplementation; Dietary supplement; Randomized clinical study

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary supplement (Active Comparator): The subjects will be instructed to take 1 tablet of either the dietary supplement or placebo twice a day, during the main meals (breakfast and lunch time), for 8 weeks
  Interventions: Dietary Supplement: Standardized Grape Seed Extract
- Placebo (Placebo Comparator): The subjects will be instructed to take 1 tablet of either the dietary supplement or placebo twice a day, during the main meals (breakfast and lunch time), for 8 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Standardized Grape Seed Extract — Grape seed dry extract standardized to provide: ≥95.0% of proanthocyanidins by spectrophotometry, ≥5.0% ≤15.0% of catechin and epicatechin by High-Performance Liquid Chromatography (HPLC)
  Arms: Dietary supplement
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate whether a standardized grape seed extract, compared to placebo, can significantly influence systolic blood pressure (SBP) in individuals with high-normal blood pressure (BP) who are adhering to a low-sodium Mediterranean diet. Additionally, the effects of the grape seed extract on diastolic blood pressure (DBP), other hemodynamic parameters, and the Perceived Stress Score will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≥18 and ≤70 years;
* Subjects with high-normal blood pressure levels, defined as SBP 130-139 mmHg and/or DBP 85-89 mmHg (according to ESH criteria);
* Subjects with an estimated 10-year CVD risk <10% (as per the SCORE risk prediction algorithm of the European Society of Cardiology);
* Subjects capable of communicating, making themselves understood, and complying with the study requirements;
* Subjects who agree to participate in the study and have dated and signed the informed consent form.

Exclusion Criteria:

* Treatment with direct vasodilator drugs or supplements known to affect blood pressure levels;
* Chronic pharmacological treatments for any clinical condition not stabilized for at least 3 months;
* Known thyroid, renal, or hepatic dysfunction (including transaminase levels ≥3 times the upper limit of normal [ULN]);
* Current or past history of alcohol abuse;
* Pregnancy or breastfeeding;
* Known intolerance or hypersensitivity to the active ingredients of the investigational dietary supplement;
* History or clinical evidence of any significant concomitant disease that could compromise subject safety or the ability to complete the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Treatment-dependent change in SBP | 8 weeks
  The primary objective is to assess and compare the effect on SBP after 8 weeks of treatment with either a standardized grape seed extract or placebo, both administered alongside a low-sodium Mediterranean diet (SOC)

SECONDARY OUTCOMES:
Treatment-dependent change in SBP | 4 weeks
  To evaluate the effect of the standardized grape seed extract on changes in SBP compared to baseline and placebo after 4 weeks of treatment
Treatment-dependent change in DBP | 4 weeks
  To evaluate the effect of the standardized grape seed extract on changes in DBP compared to baseline and placebo after 4 weeks of treatment
Treatment-dependent change in DBP | 8 weeks
  To evaluate the effect of the standardized grape seed extract on changes in DBP compared to baseline and placebo after 8 weeks of treatment
Treatment-dependent change in Augmentation Index | 8 weeks
  To evaluate the effect of the standardized grape seed extract on changes in augmentation index compared to baseline and placebo after 8 weeks of treatment
Treatment-dependent change in cfPWV | 8 weeks
  To evaluate the effect of the standardized grape seed extract on changes in the carotid-femoral pulse wave velocity (cfPWV) compared to baseline and placebo after 8 weeks of treatment
Treatment-dependent change in VOI | 8 weeks
  To evaluate the effect of the standardized grape seed extract on changes in the vascular overload index (VOI) compared to baseline and placebo after 8 weeks of treatment
Treatment-dependent change in endothelial reactivity | 8 weeks
  Change in endothelial reactivity from baseline after 8 weeks of treatment with standardized grape seed extract, compared to placebo, as assessed using the Endocheck® module integrated into the Vicorder® system.
  This method evaluates endothelium-dependent vasodilation through digital pulse volume (PV) analysis in response to reactive hyperemia. The outcome is expressed as the percent change (%) in pulse volume from baseline to peak post-occlusion values, serving as a validated surrogate marker of endothelial function.
Treatment-dependent change in arterial compliance | 8 weeks
  Change from baseline in arterial compliance, evaluated as the ratio between stroke volume (SV) and pulse pressure (PP) (SV/PP ratio), following 8 weeks of treatment with standardized grape seed extract compared to placebo.
Treatment-dependent change in the perfusion index | 8 weeks
  To evaluate the effect of the standardized grape seed extract on changes in perfusion index compared to baseline and placebo after 8 weeks of treatment
Treatment-dependent change in the perceived stress levels | 8 weeks
  Change from baseline in perceived stress levels after 8 weeks of treatment with standardized grape seed extract compared to placebo, measured using the Perceived Stress Scale (PSS) developed by Cohen and Williamson (1988).
  The PSS is a validated 10-item self-report questionnaire that assesses the degree to which situations in one's life are appraised as stressful over the past month. The questions concern the participant's feelings and thoughts during the last month. For each item, the participant indicates how often they felt or thought a certain way by circling the frequency.
  Scores range from 0 to 40, with higher scores indicating higher perceived stress levels. The outcome is expressed as the change in total PSS score from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Policlinico S.Orsola-Malpighi, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schon C, Allegrini P, Engelhart-Jentzsch K, Riva A, Petrangolini G. Grape Seed Extract Positively Modulates Blood Pressure and Perceived Stress: A Randomized, Double-Blind, Placebo-Controlled Study in Healthy Volunteers. Nutrients. 2021 Feb 17;13(2):654. doi: 10.3390/nu13020654. PMID 33671310
- [Background] Hasbal-Celikok G, Kara M, Sanchez M, Owsianik C, Gomez-Serranillos P, Yilmaz-Ozden T, Oztas E, Zengin OS, Ozhan G, Arda N, Tunc M, Sahin S, Shafiq A, Kanwal A, Ujjan HI, Rabbani F, Petrangolini G, Khan A. In Vitro Mechanistic Studies of a Standardized Sustainable Grape Seed Extract for Potential Application as a Mood-Modulating and Cognition-Enhancing Supplement. Nutrients. 2024 Oct 12;16(20):3459. doi: 10.3390/nu16203459. PMID 39458455
- [Background] Belcaro G, Ledda A, Hu S, Cesarone MR, Feragalli B, Dugall M. Grape seed procyanidins in pre- and mild hypertension: a registry study. Evid Based Complement Alternat Med. 2013;2013:313142. doi: 10.1155/2013/313142. Epub 2013 Sep 19. PMID 24171039